CLINICAL TRIAL: NCT01390623
Title: Efficacy and Safety Study of Short Term Antibiotic During Seven Days With Ceftriaxone Intravenous the First Day Then Cefixime the Second Day Till the Seventh Day of Acute Uncomplicated Pyelonephritis in Women Between 18 and 65 Years Old
Brief Title: Efficacy and Safety Study of Short-term Antibiotic for Pyelonephritis in Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0098; 2010-023697-39 (EudraCT Number)
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Acute Uncomplicated Pyelonephritis
Keywords: Acute Uncomplicated Pyelonephritis; Short-term antibiotic; Ceftriaxone; Cefixime; Women; Efficacy
MeSH Terms: interventions — Ceftriaxone

INTERVENTIONS:
Drug: Ceftriaxone — Patients will be included by investigators or coinvestigateurs, the day of consultation in the emergency adult department in Clermont-Ferrand city.
  The diagnosis of acute uncomplicated pyelonephritis is established in the emergency department based on the clinical, laboratory and imaging criteria.

SUMMARY:
Urinary tract community infections are one of very frequent reason consultation and prescription. Urinary tract represents the second site of bacterial community infection after the respiratory system. The management of the acute uncomplicated pyelonephritis was simply codified in the past recommendations of the French Agency for Safety Health Products (AFSSAPS) in 2008. Treatment is based on two main families of antibiotics, fluoroquinolones with 7 days treatment and 3rd generation cephalosporins with 10 to 14 days treatment.

The practice of a short treatment with ceftriaxone intra venous relayed by cefixime orally provides a simplified treatment for patients, a reduced use of fluoroquinolones and a probable decrease in correlation with the emergence of fluoroquinolones resistance, and finally, a decrease in the cost of treatment of acute uncomplicated pyelonephritis.

DETAILED DESCRIPTION:
Patients will be included by investigators or coinvestigateurs, the day of consultation in the emergency adult department in Clermont-Ferrand city.

The diagnosis of acute uncomplicated pyelonephritis is established in the emergency department based on the clinical, laboratory and imaging criteria.

Clinical, biological and radiological data will gathered during this consultation :

* Clinical data: flank pain, fever, urinary symptoms,
* Biological data: urine dipstick (BU No. 1), cytobacteriological urinary (ECBU No. 1), blood prélèvements (Blood count, creatinine, CRP)
* Imagery: renal and bladder ultrasound. During the next consultations in the emergency department, respectively on day 3 (J3) of treatment and on day 9 (J9), urine tests (urinary dipsticks [BU No. 2 and No. 3] and cytobacteriological urinary [ECBU No. 2 and No. 3] will be realised. The clinical and biological management of patient will be performed by the same department to ensure a better comparability of biological results and a centralized real-time clinical data.

Patient follow-up will end with a phone call on day 37 (J37), and the rate of clinical relapses and / or biological occurred between day 9 and day 37.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 65 years old
* Diagnosis of Acute Uncomplicated Pyelonephritis
* Patient obliged to participate in the French national health and pensions system.
* Patient who have read, understood and signed the consent

Exclusion Criteria:

* Women who are pregnant
* Men
* One of these risk factor who define a complicated pyelonephritis:

Medical history of uro-nephrology problem Nephropathy Obstructive Uropathy Vesicoureteral reflux Post mictinal residue > 100mL Urinary fistula Catheter vesicle and urethral Kidney transplantation Immunodeficiency Diabetes

* Recurrent pyelonephritis
* Allergy of betalactam or cephalosporin
* History of hypersensitivity reactions to antibiotic medications
* Patient in terminal care
* Trouble of cognitive function
* Patient deprive of judicial or administrative freedom
* Patient participating to another trial
* Refusal to participate to the trial

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-07; Primary Completion 2013-07 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Microbiological cure at the 9th day | at the 9th day

SECONDARY OUTCOMES:
Microbiological cure at the 3 rd day | at the 3 rd day
Number of recurrence of acute pyelonephritis during the month after the treatment between the 9 th and the 37 th day | between the 9 th and the 37 th day

CONTACTS AND LOCATIONS:
Overall Officials: Thierry MATHEVON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moustafa F, Nguyen G, Mathevon T, Baud O, Saint-Denis J, Dublanchet N, Pereira B, Shinjo C, Romaszko JP, Dopeux L, Dutheil F, Schmidt J. Evaluation of the efficacy and tolerance of a short 7 day third-generation cephalosporin treatment in the management of acute pyelonephritis in young women in the emergency department. J Antimicrob Chemother. 2016 Jun;71(6):1660-4. doi: 10.1093/jac/dkw021. Epub 2016 Feb 21. PMID 26903277